CLINICAL TRIAL: NCT05931653
Title: Multimodal Physical Therapy Approach With and Without Proprioceptive Training in Lumber Facet Joint Syndrome.
Brief Title: Multimodal PT With and Without Proprioceptive Training in Lumber FJS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/1102
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Facet Joint Pain
Keywords: Low back pain; Facet joint; Range of motion; Balance; Fatigue; Lordosis
MeSH Terms: conditions — Low Back Pain; Fatigue; Lordosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal Physical Therapy (Experimental): Multimodal Physical therapy/Traditional Physical therapy
  Interventions: Other: Multimodal Physical therapy
- Proprioceptive training along with Multimodal Physical Therapy (Experimental): Proprioceptive training along with Multimodal Physical Therapy
  Interventions: Other: Proprioceptive training along with and Multimodal Physical therapy

INTERVENTIONS:
Other: Multimodal Physical therapy — • Multimodal Physical therapy: Hot pack for 15 mins, TENS for 15 mins, Ultrasound at 1.5 W/cm2 intensity for 5 mins, Soft tissue release for <5-15 mins as per need, HVLA, PA Glides (Central and Transverse mobilizations) (10 sec each) x5 sets, Lumbar facet gapping (LFG) in side lying (10 sec 3 sets) and Lumbar rotational facet gapping (LRFG) in side lying (10 sec 3 sets). 03 days/week for 06 weeks.
  Arms: Multimodal Physical Therapy
Other: Proprioceptive training along with and Multimodal Physical therapy — * Multimodal Physical Therapy: Hot pack-5 mins, TENS-5 mins, U.S (1.5 W/cm2)-5 mins, Soft tissue release-<5-15 mins, HVLA, PA Glides (Central and Transverse)-10 sec each 5 sets, Lumbar facet gapping-10 sec 3 sets and Lumbar rotational facet gapping-10 sec 3 sets. 3 days/week for 6 weeks.
  * Proprioceptive Training:1. Trunk Balance (15 mins). In sitting, kneeling, quadruped, and supine positions for 30 seconds to 2 minutes. Progression to more challenging. Each will be performed for 2-3 mins. In case of pain exercise will be interrupted and substituted with another one.
    2. PNF Training (10-12 mins). Each PNF training-1 set of 15 reps with 30s rest between and 60s after 15 reps. Week 1-2 alternate full isometrics of trunk flexors and extensors for 10s in sitting. Week 3-4, 5s resisted concentric, 5s eccentric and 5s isometrics contractions in forward and backward bending. Week 5-6, alternate chop and lift movement patterns of upper extremities in diagonal and spiral directions for 10s.
  Arms: Proprioceptive training along with Multimodal Physical Therapy

SUMMARY:
This will be a randomized clinical trial. The study will be conducted at Pakistan Railways General Hospital Rawalpindi and Riphah International Hospital Islamabad. Patients with FJS will be included. The aim of this study is to find the comparative effects of multimodal physical therapy treatment and proprioceptive training along with multimodal physical therapy treatment on pain, lumbar ranges of motion, disability, fatigue, lumbar lordosis curvature and balance.

Participants will be assessed for pain, lumbar range of motions, lumbar lordosis, disability, fatigue and balance before treatment. The intervention duration is 06 weeks, 03 sessions per week will be given to all participants. Pain and lumbar ranges of motion will be measured on every visit. At the end of 06th week final readings for functional status, fatigue level, lumbar lordosis angle, fall risk and limits of stability will also be recorded. Data will be analyzed by SPSS v.23.

ELIGIBILITY:
Inclusion Criteria:

* Patients with facet joint syndrome diagnosed by standard criteria. This criterion includes:

  * One point tenderness under X-ray radiography
  * Kemp sign.
  * Catching pain.
  * Pain increases with lumbar extension.
  * Pain with bilateral SLR.
  * Or pain diminishes with Medial branch block or Facet joint block.
  * Provocation Maneuver. Acevedo sign (Facet stress sign) Unilateral facet palpation Percussion spinal test Impaired range of motion Jump test
  * Revel's criteria 05 out of 07- 1. age greater than 65 years and pain that was not exacerbated by coughing, not worsened by hyperextension, not worsened by forward flexion, not worsened when rising from flexion, not worsened by extension-rotation, and well-relieved by recumbency.

Standing flexion, returning from standing flexion, standing extension, the extension rotation test.

* On Biodex balance system (BBS), overall stability index between 0.7-2.8.
* On Biodex balance system (BBS) Limits of stability Anterior: less than 80, posterior: less than 40 and lateral: less than 160 (80 on each side) 75% LOS (moderate level).
* NPRS ratings greater than 4
* Constant or Intermittent pain worsening on repeated movements

Exclusion Criteria:

* T-score of -2.5 or lower.
* BMI is 30.0 or higher.
* Patients with Lumbar Postural Syndrome
* Patients with Lumbar Instability
* Post laminectomy/discectomy
* Spondylolisthesis
* Osteoporosis/Fractures
* Cauda equine syndrome
* Recent history of spinal trauma or surgery
* Lumbar myelopathy
* Patients with known metabolic diseases
* Participants having less than 20% ODI scoring

Ages: 25 Years to 53 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 6th week
  Changes from base Line Visual Analogue Rating (VAS) is a self-report of clinical pain intensity. The scale was 10 cm long and anchored by the statements "no pain" (0-4 mm) on the left mild pain (5-44 mm), moderate pain (45-74 mm), and the most intense pain imaginable (75-100 mm) on the right.
Bubble Inclinometer | 6th week
  Changes from base Line Bubble inclinometers assess range of motion like a goniometer. The 12th thoracic and 1st sacral vertebrae will be taken as the reference points for lumbar flexion and extension.
Lateral view X-ray and Kinovea software | 6th week
  Changes from base Line Angle of lumbar lordosis will be measures by plane X-ray lateral view and angle will be measured by Kinovea software for windows platform.
Modified Oswestry Disability Index (MODI) Urdu Version | 6th week
  Changes from base Line MODI is a measure of disability in low back pain. It is divided into ten sections that assess the level of pain and interference with physical activities such as sleeping, standing, walking, home making, social life and traveling. Each question has a possible six responses which are scored from 0 to 5. The score for each section is added and divided by the total possible score (fifty if all sections are completed), with the resulting score multiplied by a hundred to yield a percentage score with 0% equivalent to no disability and 100% equivalent to a great deal of disability.
Limits of stability by Biodex Balance System (BBS) | 6th week
  Changes from base Line In testing mode of BBS Score be calculated at moderate difficulty level (75%-default set value). This test challenges patients to move and control their center of gravity within their base of support. Patients must shift their weight to move the cursor from the center target to a blinking target and back as quickly and with as little deviation as possible. The same process is repeated for each of nine targets. Targets on the screen blink in random order.
Fall Risk Scoring by Biodex Balance System (BBS) | 6th week
  Changes from base Line Normal actual score range of fall risk index for individuals ranging 17 to 53 years of age is 0.7 to 2.8. The closer an individual to this actual core range, he/she is considered more stable with reduction in fall risk.
Fatigue by Fatigue Assessment Scale (FAS) | 6th week
  Changes from base Line Every point of the fatigue assessment scale has further five components in which 1 means "never" and 5 means "always" Its scoring is from 10-50 in which 10 showing lowest fatigue level and 50 means indicating highest fatigue level. The fatigue assessment scale total count can be obtained by adding the numbers obtained of the queries altogether. If the overall score is less than 22 it denotes no fatigue, more than 22 it will show fatigue. 10-21 Score of FAS: fatigue is not present. 22-50 score of FAS: the presence of substantial fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Affan Iqbal, PhD*, Principal Investigator — Riphah College of Rehabilitation and Allied Health Sciences, Riphah International University; Syed A Shakil-Ur-Rehman, PhD, Study Chair — Riphah College of Rehabilitation and Allied Health Sciences, Riphah International University
Locations (3):
- Pakistan (3):
  - Riphah Rehabilitation Center, Rawalpindi, Punjab Province
  - Pakistan Railways General Hospital, Rawalpindi, Punjab Province
  - The Health Professionals, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No